CLINICAL TRIAL: NCT07408024
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase IIa Clinical Study to Evaluate the Efficacy and Safety of TollB-001 Tablets in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: Study of TollB-001 Tablets in Moderate to Severe Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Toll Biotech Co. Ltd. (Beijing) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLBT-TOLLB-001-IIa; CTR20253314 (Other: CDE)
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TollB-001 (Experimental)
  Interventions: Drug: Group 1: TollB-001 100mg qd po; Group 2: TollB-001 200mg qd po; Group 3: TollB-001400mg qd po
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Group 1: TollB-001 100mg qd po; Group 2: TollB-001 200mg qd po; Group 3: TollB-001400mg qd po — for 4 weeks
  Arms: TollB-001
Drug: Placebo — matching placebo qd po for 4 weeks
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the safety, pharmacokinetic (PK) characteristics, and preliminary efficacy of a new oral chemical drug in : adults aged 18-70 years (male or female) with moderate to severe active rheumatoid arthritis (RA), who have had inadequate response to or intolerance of at least one conventional synthetic disease-modifying antirheumatic drug (csDMARDs) .

Participants will take the assigned study drug (either tollB-001 Tablets or placebo) once daily orally for 4 weeks, follow up for 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years (inclusive) at the time of signing the informed consent form, regardless of gender.
2. Diagnosis of RA according to the 1987 American College of Rheumatology (ACR) criteria or the 2010 ACR/European League Against Rheumatism (EULAR) classification criteria.
3. DAS28-CRP > 3.2 at screening (joints that have undergone major surgical treatment or intra-articular injection of glucocorticoids or hyaluronic acid within 6 weeks before randomization are not counted in the TJC and SJC counts).
4. C-reactive protein (CRP)/high-sensitivity C-reactive protein (hsCRP) ≥ upper limit of normal (ULN) at screening.
5. Prior to the first administration of the study drug, has received continuous treatment with at least one conventional synthetic disease-modifying antirheumatic drug (csDMARDs, including methotrexate, chloroquine, hydroxychloroquine, sulfasalazine, leflunomide, iguratimod) with inadequate response or intolerance, and agrees to discontinue use during the study.
6. Female and male subjects of childbearing potential must use effective contraceptive measures during the study and for 3 months after the last study drug administration. Male subjects whose spouses or partners are females of childbearing potential must also agree to use effective contraceptive measures during the study and for 3 months after the last administration, and shall not donate sperm during this period. Female subjects of childbearing potential must have a negative pregnancy test.
7. Must provide written informed consent and be willing and able to comply with the study protocol (e.g., understand and complete questionnaires, follow the visit schedule, take medications as prescribed).

Exclusion Criteria:

1. Hypersensitivity to the study drug or any of its components.
2. ACR functional class IV or being bedridden/wheelchair-bound for a long time.
3. Use of any of the following drugs or treatments:

   Prior use of Janus kinase (JAK) inhibitors (including but not limited to tofacitinib, baricitinib, upadacitinib), biologic disease-modifying antirheumatic drugs (bDMARDs), or participation in clinical trials of the aforementioned drugs.

   Use of csDMARDs within 28 days before randomization (leflunomide within 56 days before administration, or subjects who have received standard cholestyramine treatment or activated charcoal washout within 28 days are not eligible for enrollment).

   Use of other known drugs with strong immunosuppressive or immunomodulatory effects (such as puerarin, tripterygium wilfordii, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, 6-mercaptopurine, etc.) other than the above within 4 weeks before randomization.

   Receipt of any parenteral (intramuscular or intravenous) or intra-articular glucocorticoids within 4 weeks before randomization.

   Receipt of interferon treatment within 4 weeks before randomization. Oral traditional Chinese medicine for the treatment of RA and other inflammatory diseases within 4 weeks before randomization.

   Use of opioid drugs within 1 week or 5 drug half-lives (whichever is longer) before the first administration of the study drug.

   Receipt of integrin αV antibodies or cell depletion therapy within 3 months or 5 half-lives (whichever is longer) before the screening visit.
4. History or evidence of any of the following diseases:

   Other systemic inflammatory diseases except RA (excluding secondary Sjögren's syndrome), including but not limited to juvenile chronic arthritis, Crohn's disease, ulcerative colitis, psoriatic arthritis, systemic lupus erythematosus, ankylosing spondylitis, reactive arthritis, systemic vasculitis, gout, or other joint diseases that may affect efficacy evaluation (e.g., osteoarthritis with significant joint pain).

   Felty's syndrome. Any active malignant tumor or history of malignant tumor. Chronic pain history that may affect study evaluation. Active tuberculosis, latent untreated tuberculosis, or incompletely cured tuberculosis as judged by the investigator and/or specialist.

   History of any persistent or chronic infection (e.g., chronic pyelonephritis, bronchiectasis, osteomyelitis) deemed inappropriate for study participation by the investigator, or oral anti-infective drugs (excluding onychomycosis) within 14 days before the first administration of the study drug; history of deep space/tissue infection (e.g., fasciitis, abscess, osteomyelitis) within 52 weeks before the screening visit.

   Poorly controlled severe diseases such as diabetes mellitus, hypertension, kidney disease, neurological disease, liver disease, severe heart disease (e.g., decompensated heart failure [New York Heart Association Class III or IV], unstable angina pectoris, myocardial infarction, etc.), respiratory disease, severe chronic gastrointestinal disease (e.g., active or recurrent peptic ulcer), or prior treatment that may affect drug absorption (e.g., gastrointestinal surgery) and deemed by the investigator to potentially hinder the subject's participation in the study.

   Major surgery within 8 weeks before randomization or expected to undergo major surgery after enrollment.
5. Any laboratory abnormalities meeting the following criteria at screening:

   Hemoglobin < 90.0 g/L. Total white blood cell count < 2.5 × 10⁹/L. Neutrophil count < 1.5 × 10⁹/L. Lymphopenia (lymphocyte count < 750 cells/μL). Platelet count < 100 × 10⁹/L.
6. Positive hepatitis B surface antigen (HBsAg); or positive hepatitis B core antibody (HBcAb) with HBV DNA above the lower limit of detection; positive hepatitis C virus (HCV) antibody with positive HCV-RNA; positive human immunodeficiency virus (HIV) antibody or positive syphilis antibody.
7. Drug or alcohol abuse or dependence at screening, or history of drug or alcohol abuse or dependence within 6 months before randomization.
8. Participation in any clinical trial of drugs or medical devices within 4 weeks or 5 half-lives (whichever is longer) before randomization.
9. Blood donation ≥ 400 mL or receipt of blood transfusion within 3 months before randomization.
10. Any other factors deemed by the investigator to potentially affect the conduct or result evaluation of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety-AE/lab tests/PE/VS/ECG | up to week 8
  Safety parameters including the incidence of adverse events (AEs), abnormalities in laboratory tests, physical examinations, vital signs, and routine 12-lead electrocardiograms

SECONDARY OUTCOMES:
Efficacy-ACR20 | Day8, Day15, Day29, Day56
  Proportion of patients achieving 20% improvement in the ACR RA disease activity core criteria (ACR20) at each post-baseline visit;
EfficacyACR50/70 | Day8, Day15, Day29, Day56
  Proportion of patients achieving 50% (ACR50) and 70% (ACR70) improvement at each post-baseline visit;
Efficacy-DAS28 | Day8, Day15, Day29, Day56
  Proportion of patients achieving DAS28-CRP < 2.6, DAS28-CRP ≤ 3.2, DAS28-ESR < 2.6, and DAS28-ESR ≤ 3.2 at each post-baseline visit
Efficacy-CDAI | Day8, Day15, Day29, Day56
  Changes in Clinical Disease Activity Index (CDAI) from baseline at each post-baseline visit
Efficacy-morning stiffness | Day8, Day15, Day29, Day56
  Changes in morning stiffness duration from baseline at each post-baseline visit; Assessment Time: Each post-baseline visit
Efficay-patient assessment of arthritis pain | Day8, Day15, Day29, Day56
  Changes in Patient's Assessment of Arthritis Pain (PtAAP) from baseline at each post-baseline visit
Efficacy-patient global assessment | Day8, Day15, Day29, Day56
  Changes in Patient's Global Assessment of Disease Activity (PtGA) from baseline at each post-baseline visit;
Efficacy-physician's global assessemnt | Day8, Day15, Day29, Day56
  Changes in Physician's Global Assessment of Disease Activity (PhGA) from baseline at each post-baseline visit
Efficacy-DAQ-DI | Day8, Day15, Day29, Day56
  Changes in Health Assessment Questionnaire-Disability Index (HAQ-DI) scores from baseline at each post-baseline visit
Efficay-ESR | Day8, Day15, Day29, Day56
  Changes in erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) from change in ESR from baseline at each post-baseline visit
Efficay-CRP | Day8, Day15, Day29, Day56
  Changes in C-reactive protein (CRP) from baseline at each post-baseline visit
Secondary | Up to week 4
  Serum concentration of TollB-001

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Linfen Central Hospital, Linfen, Shanxi

IPD SHARING:
Plan to Share IPD: No